CLINICAL TRIAL: NCT05307991
Title: Integrating Enhanced HIV Pre-exposure Prophylaxis Into a Sexually Transmitted Infection Clinic in Lilongwe
Brief Title: Integrating Enhanced HIV PrEP Into a STI Clinic in Lilongwe
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 21-2457
Record Dates: First submitted 2022-03-24; First posted 2022-04-01 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-04

CONDITIONS: HIV Infections; Sexually Transmitted Diseases; Blood-Borne Infections; Communicable Disease; Infections; Sexually Transmitted Diseases, Bacterial; Sexually Transmitted Diseases, Viral; RNA Virus Infections; Virus Disease; Syphilis; Neisseria Gonorrheae Infection; Chlamydia Trachomatis Infection
Keywords: Tenofovir; Pre-exposure prophylaxis; emtricitabine; assisted partner notification
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Blood-Borne Infections; Communicable Diseases; Infections; Sexually Transmitted Diseases, Bacterial; Sexually Transmitted Diseases, Viral; RNA Virus Infections; Virus Diseases; Syphilis; Gonorrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Index PrEP participants: This group includes persons 15 years and older who are started on PrEP at the STI clinic. Participants in this group will be followed for 6 months, with follow-up visits at 1, 3, and 6 months, and will be asked to refer sexual partners from the preceding 6 months as well as any new sexual partners throughout the study period. They will also receive testing for Neisseria gonorrhea, Chlamydia trachomatis, and syphilis (depending on prior results) at baseline, 3, and 6 months. A sub-group of participants will also complete in-depth interviews to contextualize observed behaviors and outcomes.
  Interventions: Drug: PrEP; Device: STI testing; Behavioral: Assisted partner notification; Diagnostic Test: Acute HIV testing
- Non-PrEP participants: This group includes persons who are eligible to receive PrEP but who decline initiation at their index visit to the STI clinic. These participants will be followed for 6 months, with follow-up visits at 3 and 6 months, and receive testing for Neisseria gonorrhea, Chlamydia trachomatis, and syphilis (depending on prior results) at baseline, 3, and 6 months. However, at any time during the follow-up period these persons can choose to initiate PrEP. This would not change their follow-up frequency nor their assigned group, and they would continue to be followed for 6 months from the date of initial enrollment. A sub-group of participants will also complete in-depth interviews to contextualize observed behaviors and outcomes.
  Interventions: Device: STI testing
- Partner participants: This group is made up of named/referred partners from the Group 1 (Index PrEP participant) who are eligible for and agree to start PrEP. They will receive identical intervention to that of the Group 1, specifically: this group will be followed for 6 months, with follow-up visits at 1, 3, and 6 months, and will be asked to refer sexual partners from the preceding 6 months as well as any new sexual partners throughout the study period. They will also receive testing for Neisseria gonorrhea, Chlamydia trachomatis, and syphilis (depending on prior results) at baseline, 3, and 6 months. A sub-group of participants will also complete in-depth interviews to contextualize observed behaviors and outcomes.
  Interventions: Drug: PrEP; Device: STI testing; Behavioral: Assisted partner notification; Diagnostic Test: Acute HIV testing
- Providers: This group is made up providers involved in the provision of PrEP or other related services including STI management, HIV testing or counseling, or assisted partner notification (aPN). Examples include: clinicians, nurses, HIV testing/aPN counselors, registration staff, community tracers, and clinic management who provide clinical or aPN services. These participants will be asked to complete a survey responding to acceptability, feasibility, and appropriateness of the enhanced PrEP implementation strategy as an integrated strategy within the STI clinic. They will also participate in in-depth interviews. These activities will be completed at baseline and approximately 6 months thereafter.

INTERVENTIONS:
Drug: PrEP — HIV pre-exposure prophylaxis (or PrEP) will include the Malawi-approved PrEP regimen at time of study enrollment. At time of submission, the only Malawi-approved regimen includes Tenofovir/emtricitabine (TDF/FTC) containing 300 mg of TDF and 200 mg of FTC. If additional PrEP regimens become available in Malawi during the study recruitment or follow-up, participants will be able to choose from any regimen that they are eligible to receive per Malawi PrEP guidelines.
  Groups: Index PrEP participants; Partner participants
Device: STI testing — Urine specimens will be tested for Chlamydia trachomatis (Ct) and Neisseria gonorrhoeae (GC) using GeneXpert® (Cepheid, Sunnyvale, CA) Xpert® CT/GC platform and cartridge and syphilis RPR titer (BD Macro-VUE™, Becton, Dickinson and Company, Franklin Lakes, NJ [FDA approved]) with confirmatory Treponema pallidum particle agglutination (TP-PA) (Serodia Fujirebio Inc, Malvern, PA [CE mark]) if RPR is positive.
  Groups: Index PrEP participants; Non-PrEP participants; Partner participants
Behavioral: Assisted partner notification — Participants will be asked to provide the name and locator information for all sexual partners in the preceding 6 months. Participants will be asked to refer sexual partners to the clinic and will be provided with cards to distribute to partners. Each card will request that the recipient report to the STI clinic with the card and will contain a linking number that links them back to the index participant.
  Sexual Partner Tracing: In accordance with the contract referral approach, if the named partners do not present to an STI clinic within 7-14 days, community outreach workers will contact the partners and counsel them to visit the clinic. Contact may be made through telephone, text message, or in person, as needed and will not disclose the name or identify of the index patient.
  Groups: Index PrEP participants; Partner participants
Diagnostic Test: Acute HIV testing — Persons initiating or re-initiating PrEP will also be screened for acute HIV infection (AHI) using Abbott RealTime HIV-1 Assay (Abbott Laboratories, Chicago, IL) or Xpert® HIV-1 Viral Load (GeneXpert, Cepheid, Sunnyvale, CA).
  Groups: Index PrEP participants; Partner participants

SUMMARY:
This is a prospective cohort study evaluating acceptability, feasibility, and effectiveness of integrating HIV pre-exposure prophylaxis (PrEP) into a sexually transmitted infection (STI) clinic alongside assisted partner notification and etiologic STI testing in Lilongwe, Malawi.

ELIGIBILITY:
Patient Participant

Inclusion Criteria:

* ≥15 years of age.
* Eligible for PrEP according to Malawi PrEP guidelines (see below)
* Presenting for care at STI clinic (primary presentation or referral from partner based on STI or HIV exposure)
* Able to consent for study participation and willing to provide locator information for follow-up tracing

  *Malawi PrEP eligibility criteria:
* Age ≥15 years
* HIV seronegative iii. At substantial risk for HIV, with prioritization of persons who:
* Buy or sell sex; Key population (female sex worker, men who have sex with other men, transgendered persons; Vulnerable population included adolescent girls and young women aged 15-24; STI clients; Serodiscordant couples including HIV-negative women who are pregnant or breast feeding or HIV-negative men or women for whom their HIV-infected partner is: not on ART, on ART <6 months, has an unsuppressed or high viral load, or is non-adherent to ART, iv. Have ruled out acute HIV infection, or defer PrEP initiation for anyone with signs or symptoms consistent with acute HIV infection, v. Willingness to attend scheduled PrEP visits, vi. No contraindication to use of TDF and 3TC, vii. Bodyweight ≥30 kg, viii. Estimated glomerular filtration rate (eGFR) ≥60mL/min, ix. No known renal diseases, x. No diabetes mellitus.

Exclusion Criteria:

* Current imprisonment or incarceration in a medical or psychiatric facility

Provider Participant:

Inclusion Criteria:

* ≥18 years of age.
* Duties relevant to integration or provision of PrEP and/or aPN at STI clinic

Exclusion Criteria:

- Unable or unwilling to provide informed consent

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patient participants are PrEP-eligible persons who are seeking care in an STI clinic in Lilongwe, Malawi, including sexual partners who are referred by index participants and initiated on PrEP.
  Provider participants include persons who are involved in aspects of patient care that includes: screening for, prescribing, or managing PrEP; eliciting or tracing sexual partners; counseling STI clinic patients on HIV risk and risk reduction. Examples include: clinicians, nurses, HIV testing/aPN counselors, registration staff, community tracers, and clinic management who provide clinical or aPN services.
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Proportion of participants retained on PrEP | Approximately 6 months after enrollment
  Examine the proportion of participants who initiate PrEP at enrollment who are retained on PrEP through study completion (6 months)
Number of participants retained on PrEP | Approximately 6 months after enrollment
  Examine the number of participants who initiate PrEP at enrollment who are retained on PrEP through study completion (6 months)
Number of provider participants describing feasibility of aPN and STI testing (qualitative) | Approximately 6 months after the start of enrollment
  To gain deeper insights about the feasibility of enhanced PrEP delivery, PrEP providers from the study site will be asked to participate in in-depth interviews. Participating providers are involved in different aspects of PrEP provision, aPN, and STI testing and include study staff members. Feasibility is defined as a positive rating about the intervention's potential performance in real-life conditions at the clinic and community levels.
Number of provider participants describing feasibility of aPN and STI testing (quantitative) | Approximately 6 months after the start of enrollment
  To gain deeper insights about the feasibility of enhanced PrEP delivery, PrEP providers from the study site will be asked to complete survey using modified validated measures assessing feasibility on a 5-point Likert scale. Participating providers are involved in different aspects of PrEP provision, aPN, and STI testing and include study staff members.
Number of provider participants describing acceptability of aPN and STI testing (quantitative) | Approximately 6 months after the start of enrollment
  To gain deeper insights about the acceptability of enhanced PrEP delivery, PrEP providers from the study site will be asked to complete survey using modified validated measures assessing feasibility on a 5-point Likert scale. Participating providers are involved in different aspects of PrEP provision, aPN, and STI testing and include study staff members.
Number of provider participants describing acceptability of aPN and STI testing (qualitative) | Approximately 6 months after the start of enrollment
  To gain deeper insights about the acceptability of enhanced PrEP delivery, PrEP providers from the study site will be asked to participate in in-depth interviews. Participating providers are involved in different aspects of PrEP provision, aPN, and STI testing and include study staff members. Acceptability is defined as a positive rating about the intervention's potential performance in real-life conditions at the clinic and community levels.
Number of patient participants describing acceptability of aPN and STI testing (qualitative) | Approximately 6 months after enrollment
  To gain deeper insights about the acceptability of enhanced PrEP delivery from the patient perspective, as subset of enrolled patients (including persons who initiate PrEP [index], referred partners who initiate PrEP, and persons who decline PrEP) will be asked to participate in in-depth interviews. Acceptability is defined as a positive rating about the intervention's potential performance in real-life conditions at the clinic and community levels.
Number of patient participants describing acceptability of aPN and STI testing (quantitative) | Approximately 6 months after enrollment
  To gain deeper insights about the acceptability of enhanced PrEP delivery from the patient perspective, participants will be asked a series of questions using modified validated measures assessing acceptability on a 4-point Liker scale. Acceptability is defined as a positive rating about the intervention's appeal.
Number of patient participants describing feasibility of aPN and STI testing (qualitative) | Approximately 6 months after enrollment
  To gain deeper insights about the feasibility of enhanced PrEP delivery from the patient perspective, as subset of enrolled patients (including persons who initiate PrEP [index], referred partners who initiate PrEP, and persons who decline PrEP) will be asked to participate in in-depth interviews. Acceptability is defined as a positive rating about the intervention's potential performance in real-life conditions at the clinic and community levels.

SECONDARY OUTCOMES:
Number of STI clinic patients eligible for PrEP | Approximately 1 year
  The number of STI clinic patients who would meet Malawi PrEP eligibility according to pre-defined criteria
Proportion of STI clinic patients eligible for PrEP | Approximately 1 year
  The proportion of STI clinic patients who would meet Malawi PrEP eligibility
Number of PrEP eligible STI clinic patients referred for PrEP | Approximately 1 year
  The number of PrEP eligible STI clinic patients who are referred for PrEP services
Proportion of PrEP eligible STI clinic patients referred for PrEP | Approximately 1 year
  The proportion of PrEP eligible STI clinic patients who are referred for PrEP services
Number of PrEP eligible STI clinic patients declining PrEP | Approximately 1 year
  Reasons for declining PrEP will be reported qualitatively in order to inform future studies.
Number of PrEP-eligible patients starting PrEP within 7-days of STI screening | Approximately 1 year
  The number of PrEP-eligible patients starting PrEP within 7-days of presenting for initial STI screening
Proportion of PrEP-eligible patients starting PrEP within 7-days of STI screening | Approximately 1 year
  The proportion of PrEP-eligible patients starting PrEP within 7-days of presenting for initial STI screening
Proportion of all participants retained on PrEP | Up to approximately 6 months
  The proportion of participants (including persons who initiate PrEP [index], referred partners who initiate PrEP, and persons who initially decline PrEP but start during study follow-up) who are retained on PrEP at 1, 3, and 6 months of follow-up.
Proportion of enrolled PrEP users naming at least one recent sex partner | Up to approximately 6 months
  The proportion of PrEP users who name at least one recent sex partner, defined as having had sex with them in the prior 6 months, for assisted partner notification
Number of named partners screened for PrEP eligibility | Approximately 1 year
  The number of named partners who return for PrEP screening using either passive notification or those who return only after tracing
Proportion of named partners screened for PrEP eligibility | Approximately 1 year
  The proportion of named partners who return for PrEP screening using either passive notification or those who return only after tracing
Number of named partners screened for PrEP eligibility who are ineligible for PrEP | Approximately 1 year
  Among partners presenting for screening, the number of named partners who are ineligible for PrEP.
Proportion of named partners screened for PrEP eligibility who are ineligible for PrEP | Approximately 1 year
  Among partners presenting for screening, the proportion of named partners who are ineligible for PrEP.
Number of PrEP-eligible named partners who initiate PrEP | Approximately 1 year
  Among PrEP-eligible partners who present to the clinic, the number who agree to initiate PrEP
Proportion of PrEP-eligible named partners who initiate PrEP | Approximately 1 year
  Among PrEP-eligible partners who present to the clinic, the proportion who agree to initiate PrEP
Number of PrEP-eligible named partners who decline PrEP | Approximately 1 year
  Reasons for declining PrEP will be reported qualitatively in order to inform future studies.
Proportion of consenting eligible patient participants who receive STI testing | Up to approximately 6 months
  The proportion of all participants who receive STI testing at baseline, 0, 3, and 6 months
Proportion of participants who receive appropriate STI treatment within 7 days of testing | Up to approximately 6 months
  The proportion of all patient participants who receive indicated treatment, based on results of etiologic STI testing, within 7 days of having been tested
Proportion of participants with symptomatic STI | Up to approximately 6 months
  The proportion of all patient participants (including persons who initiate PrEP [index], referred partners who initiate PrEP, and persons who initially decline PrEP) who have a symptomatic STI at enrollment, 1, 3, or 6 months
Proportion of participants with asymptomatic STI | Up to approximately 6 months
  The proportion of all patient participants (including persons who initiate PrEP [index], referred partners who initiate PrEP, and persons who initially decline PrEP) who have an asymptomatic STI at enrollment, 1, 3, or 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Rutstein, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Bwaila STI clinic, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: beginning 9 months following publication and continuing for 36 months
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data sharing agreement with UNC.

REFERENCES:
- [Derived] Munthali T, Masano A, Chen JS, Kumwenda W, Pedersen C, Chinthenga K, Jere E, Mathiya E, Ndalama B, Nyirenda N, Bonongwe N, Chagomerana MB, Hosseinipour MC, Hoffman IF, Matoga M, Rutstein SE. Assisted partner notification as a strategy to enhance Pre-Exposure Prophylaxis (PrEP) screening and uptake - results from a prospective cohort study in Lilongwe, Malawi. BMC Health Serv Res. 2025 Jul 2;25(1):890. doi: 10.1186/s12913-025-13038-4. PMID 40604850
- [Derived] Rutstein SE, Chen JS, Jere E, Limarzi-Klyn L, Mphande Z, Mathiya E, Nyirenda N, Banda G, Mulholland GE, Hosseinipour MC, Hoffman IF, Matoga M. High Incidence of Curable Sexually Transmitted Infections Among Persons Accessing Oral Preexposure Prophylaxis at an Integrated Sexually Transmitted Infection/Preexposure Prophylaxis Clinic in Lilongwe, Malawi. Sex Transm Dis. 2025 Sep 1;52(9):577-584. doi: 10.1097/OLQ.0000000000002170. Epub 2025 Apr 22. PMID 40261957
- [Derived] Rutstein SE, Matoga M, Chen JS, Mathiya E, Ndalama B, Nyirenda N, Bonongwe N, Chithambo S, Chagomerana M, Tegha G, Hosseinipour MC, Herce ME, Jere E, Krysiak RG, Hoffman IF. Integrating Enhanced HIV Pre-exposure Prophylaxis Into a Sexually Transmitted Infection Clinic in Lilongwe: Protocol for a Prospective Cohort Study. JMIR Res Protoc. 2022 Dec 5;11(12):e37395. doi: 10.2196/37395. PMID 36469400